CLINICAL TRIAL: NCT02162420
Title: Hematopoietic Stem Cell Transplant for Dyskeratosis Congenita or Severe Aplastic Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013OC127; MT2013-34C (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Dyskeratosis Congenita; Aplastic Anemia
Keywords: severe aplastic anemia; Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Dyskeratosis Congenita; Anemia, Aplastic | interventions — Alemtuzumab; fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Stem Cell Transplantation; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm A Dyskeratosis Congenita (DKC) (non-haploidentical donor) (Experimental): Fludarabine based preparative regimen, including alemtuzumab, cyclophosphamide, fludarabine, followed by stem cell transplant for the treatment of dyskeratosis congenita.
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Stem Cell Transplant
- Arm B: Severe Aplastic Anemia (SAA ) (non-matched related, non-haploidentical donor) (Experimental): Fludarabine based preparative regimen which includes: cyclophosphamide, fludarabine, rabbit ATG and total body irradiation. Followed by stem cell transplant.
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Biological: Stem Cell Transplant; Drug: Anti-thymocyte globulin
- Arm C: Severe Aplastic Anemia (matched related donor) (Experimental): Fludarabine based preparative regimen which includes: cyclophosphamide, fludarabine, rabbit ATG and total body irradiation. Followed by stem cell transplant.
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Biological: Stem Cell Transplant; Drug: Anti-thymocyte globulin
- Arm D: Dyskeratosis Congenita (DKC), PTCy platform (Experimental): Fludarabine based preparative regimen, including alemtuzumab, cyclophosphamide, fludarabine, followed by stem cell transplant for the treatment of dyskeratosis congenita.
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Stem Cell Transplant
- Arm E: Severe Aplastic Anemia (SAA), PTCy platform (Experimental): Fludarabine based preparative regimen which includes: cyclophosphamide, fludarabine, rabbit ATG and total body irradiation. Followed by stem cell transplant.
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Biological: Stem Cell Transplant; Drug: Anti-thymocyte globulin

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab 0.2 mg/kg IV over 2 hours on days -10 to -6 from transplant.
Drug: Fludarabine — Fludarabine 40 mg/m2 IV over 1 hour on days -6 to -2 from transplant.
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide 50 mg/kg IV over 2 hours on day -7 from transplant.
Radiation: Total Body Irradiation — TBI 200 cGy as a single fraction on day -1 from transplant.
  Other Names: TBI
  Arms: Arm B: Severe Aplastic Anemia (SAA ) (non-matched related, non-haploidentical donor); Arm C: Severe Aplastic Anemia (matched related donor); Arm E: Severe Aplastic Anemia (SAA), PTCy platform
Biological: Stem Cell Transplant — Stem cell transplant on day 0.
  Other Names: HSCT
Drug: Anti-thymocyte globulin — ATG (Thymoglobulin - Rabbit ) 3 mg/kg IV on days -5 to -3 from stem cell transplant.
  Other Names: Rabbit ATG
  Arms: Arm B: Severe Aplastic Anemia (SAA ) (non-matched related, non-haploidentical donor); Arm C: Severe Aplastic Anemia (matched related donor); Arm E: Severe Aplastic Anemia (SAA), PTCy platform

SUMMARY:
Fludarabine-based preparative regimen followed by an allogeneic hematopoietic stem cell transplant using related or unrelated donor in persons 0-70 years of age diagnosed with dyskeratosis congenita or severe aplastic anemia who have bone marrow failure characterized by a requirement for red blood cell and platelet transfusions. Three different preparative regimens are included based on disease and donor type.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0 - 70 years
* Acceptable hematopoeitic stem cell donor
* Dyskeratosis Congenita (DC) with evidence of BM failure defined as:

  * requirement for red blood cell and/or platelet transfusions or
  * requirement for G-CSF or GM-CSF or erythropoietin or
  * refractory cytopenias having one of the following three

    * platelets <50,000/uL or transfusion dependent
    * absolute neutrophil count <500/uL without hematopoietic growth factor support
    * hemoglobin <9g/uL or transfusion dependent
* Diagnosis of DC with a triad of mucocutaneous features:

  * oral leukoplakia
  * nail dystrophy
  * abnormal reticular skin hyperpigmentation, or
* Diagnosis of DC with one of the following:

  * short telomeres (under a research study)
  * mutation in telomerase holoenzyme (DKC1, TERT, TERC, NOP10, NHP2, TCAB1)
  * mutation in shelterin complex (TINF2)
  * mutation in telomere-capping complex (CTC1)
* Severe Aplastic Anemia (SAA) primary transplant with evidence of BM failure:

  * Refractory cytopenia defined by bone marrow cellularity <50% (with < 30% residual hematopoietic cells)
* Diagnosis of SAA with refractory cytopenias having one of the following three:

  * platelets <20,000/uL or transfusion dependent
  * absolute neutrophil count <500/uL without hematopoietic growth factor support
  * absolute reticulocyte count <20,000/uL
* Severe Aplastic Anemia (SAA) requiring a 2nd transplant

  * Graft failure as defined by blood/marrow chimerism of < 5%
* Early myelodysplastic features
* With or without clonal cytogenetic abnormalities
* Adequate organ function defined as:

  * cardiac: left ventricular ejection fraction ≥ 35% with no evidence of decompensated heart failure
  * pulmonary: DLCO ≥30% predicted, no supplemental oxygen requirement
  * renal: Glomerular filtration rate (GFR) ≥30% predicted
* Voluntary written consent

Exclusion Criteria:

* Acute hepatitis or evidence of moderate or severe portal fibrosis or cirrhosis on biopsy
* Pregnant or lactating
* Uncontrolled infection
* Prior radiation therapy (applies to SAA patients only)
* Diagnosis of Fanconi anemia based on DEB
* Diagnosis of dyskeratosis congenita with advanced MDS or acute myeloid leukemia with >30% blasts

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor: Arm A Dyskeratosis Congenita (DKC) (non-haploidentical donor)
- Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor: Arm B: Severe Aplastic Anemia (SAA ) (non-matched related, non-haploidentical donor)
- Arm C: Severe Aplastic Anemia, Matched Related Donor: Arm C: Severe Aplastic Anemia (matched related donor)
- Arm D: Dyskeratosis Congenita, PTCy Platform: Arm D: Dyskeratosis Congenita (DKC), PTCy platform
- Arm E: Severe Aplastic Anemia, PTCy Platform: Arm E: Severe Aplastic Anemia (SAA), PTCy platform
Period: Overall Study
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm D: Dyskeratosis Congenita, PTCy Platform | Arm E: Severe Aplastic Anemia, PTCy Platform
Started | 12 | 18 | 23 | 0 | 8
Completed | 11 | 15 | 22 | 0 | 8
Not Completed | 1 | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants accrued to Arm D: Dyskeratosis Congenita, Haploidentical Donor.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm D: Dyskeratosis Congenita, PTCy Platform | Arm E: Severe Aplastic Anemia, PTCy Platform | Total
Number analyzed (Participants) | 12 | 18 | 23 | 0 | 8 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 15 | 13 | 0 | 4 | 41
  Between 18 and 65 years | 2 | 2 | 9 | 0 | 4 | 17
  >=65 years | 1 | 1 | 1 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 10 | 0 | 2 | 29
  Male | 6 | 7 | 13 | 0 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 17 | 21 | 0 | 7 | 56
  Unknown or Not Reported | 0 | 1 | 2 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 0 | 0 | 3
  Asian | 2 | 1 | 3 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 3 | 3
  White | 8 | 13 | 14 | 0 | 1 | 36
  More than one race | 0 | 0 | 3 | 0 | 2 | 5
  Unknown or Not Reported | 1 | 2 | 3 | 0 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 12 | 18 | 23 |  | 8 | 61

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Neutrophil Engraftment
Description: Incidence of neutrophil engraftment by day 42.
Time Frame: Day 42
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm E: Severe Aplastic Anemia, PTCy Platform
Number analyzed (Participants) | 12 | 18 | 23 | 8
Percentage of participants | 100 [0 to 100] | 100 [0 to 100] | 96 [82 to 100] | 100 [0 to 100]

2. Primary Outcome: Incidence of Platelet Engraftment
Description: Incidence of platelet engraftment at 1 year
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Arm E: Severe Aplastic Anemia, Haploidentical Donor: Arm E: Severe Aplastic Anemia (SAA), Haploidentical Donor
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm E: Severe Aplastic Anemia, Haploidentical Donor
Number analyzed (Participants) | 12 | 18 | 23 | 8
Percentage of participants | 100 [0 to 100] | 100 [0 to 100] | 96 [82 to 100] | 100 [0 to 100]

3. Secondary Outcome: Incidence of Regimen Related Mortality
Description: Incidence of regimen related mortality by day 100.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm E: Severe Aplastic Anemia, PTCy Platform
Number analyzed (Participants) | 12 | 18 | 23 | 8
Percentage of participants | 0 [0 to 0] | 6 [1 to 33] | 6 [1 to 33] | 0 [0 to 0]

4. Secondary Outcome: Incidence of Acute Graft-versus-host Disease
Description: Incidence of acute graft-versus-host disease by day 100.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm E: Severe Aplastic Anemia, PTCy Platform
Number analyzed (Participants) | 12 | 18 | 23 | 8
Percentage of participants | 0 [0 to 0] | 11 [0 to 25] | 9 [0 to 21] | 0 [0 to 0]

5. Secondary Outcome: Incidence of Chronic Graft-versus-host Disease
Description: Incidence of chronic graft-versus-host disease by 6 months
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm E: Severe Aplastic Anemia, PTCy Platform
Number analyzed (Participants) | 12 | 18 | 23 | 8
Percentage of participants | 0 [0 to 0] | 6 [0 to 16] | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Incidence of Chronic Graft-versus-host Disease
Description: Incidence of chronic graft-versus-host disease by 1 year
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm E: Severe Aplastic Anemia, PTCy Platform
Number analyzed (Participants) | 12 | 18 | 23 | 8
Percentage of participants | 0 [0 to 0] | 6 [0 to 16] | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Incidence of Secondary Malignancies
Description: Incidence of secondary malingancies
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm E: Severe Aplastic Anemia, PTCy Platform
Number analyzed (Participants) | 12 | 18 | 23 | 8
Percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse event and serious adverse event reporting is focused on protocol related endpoint data, as well as risks associated with research data collection.
  Protocol related endpoint data includes:
  * neutrophil engraftment and platelet engraftment
  * regimen related morality
  * acute GVHD at
  * chronic GVHD at
  * secondary malignancies
  There were no reportable adverse events in regards to research data collection (e.g. breach in confidentiality, etc.).
Groups:
- Arm E: Severe Aplastic Anemia, PTCy Platform: Arm E: Severe Aplastic Anemia (SAA),PTCy platform
Arm/Group | Arm A: Dyskeratosis Congenita, Non-Haploidentical Donor | Arm B: Severe Aplastic Anemia, Non-Matched Related, Non-Haploidentical Donor | Arm C: Severe Aplastic Anemia, Matched Related Donor | Arm D: Dyskeratosis Congenita, PTCy Platform | Arm E: Severe Aplastic Anemia, PTCy Platform
All-Cause Mortality (participants affected / at risk) | 1/12 | 3/18 | 1/23 | 0/0 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/18 | 0/23 | 0/0 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/18 | 0/23 | 0/0 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02162420/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT02162420/ICF_001.pdf